CLINICAL TRIAL: NCT00008554
Title: A Phase III, Randomised, Multicenter, Parallel, Open-Label Study to Compare the Efficacy, Safety, and Tolerability of GW433908 (1400 Mg Bid) and Nelfinavir (1250 Mg Bid) Over 48 Weeks in Antiretroviral Therapy Naive HIV-1 Infected Adults
Brief Title: Comparison of GW433908 and Nelfinavir in HIV Patients Who Have Not Had Antiretroviral Therapy
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Glaxo Wellcome (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Model: Parallel | Purpose: Treatment
Other Study IDs: 316A; APV30001
Record Dates: First submitted 2001-01-13; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2001-07

CONDITIONS: HIV Infections
Keywords: HIV-1; Drug Therapy, Combination; HIV Protease Inhibitors; Lamivudine; Nelfinavir; Reverse Transcriptase Inhibitors; Anti-HIV Agents; abacavir
MeSH Terms: conditions — HIV Infections | interventions — abacavir; Nelfinavir; Lamivudine; fosamprenavir

INTERVENTIONS:
Drug: Abacavir sulfate
Drug: Nelfinavir mesylate
Drug: Lamivudine
Drug: GW433908

SUMMARY:
The purpose of this study is to compare GW433908 and nelfinavir when each is given with abacavir and lamivudine to HIV patients who have not taken antiretroviral drugs.

DETAILED DESCRIPTION:
Patients are randomized in a 2:1 scheme to 1 of 2 treatment groups. Group 1 receives GW433908 plus abacavir (ABC) plus lamivudine (3TC); Group 2 receives nelfinavir (NFV) plus ABC plus 3TC. Patients undergo safety and efficacy assessments at the Screening Visit, Day 1 (Entry), and Weeks 1, 2, 4, 8, 12, 16, 20, 24, and every 8 weeks thereafter. A follow-up visit is performed 4 weeks after the permanent discontinuation of study drug. Detailed assessments for the development of lipodystrophy/fat redistribution occur at Day 1, Week 24, Week 48, and every 16 weeks thereafter. Patients have examinations and laboratory tests performed at visits.

ELIGIBILITY:
Inclusion Criteria

Patients may be eligible for this study if they:

* Are at least 13 years old (consent of parent or guardian required if under 18).
* Agree to use a proven barrier method of birth control (e.g., spermicide plus condom) during the study period (hormonal birth control will not be accepted), if able to have children.
* Have received less than 4 weeks treatment with any nucleoside reverse transcriptase inhibitor (NRTI) and have never received any nonnucleoside reverse transcriptase inhibitor (NNRT) or protease inhibitor (PI).
* Have a viral load (amount of HIV in the blood) of 5,000 copies/ml or more, or have a positive result at the screening visit.

Exclusion Criteria

Patients will not be eligible for this study if they:

* Abuse drugs or alcohol in a way that would interfere with the study, in the opinion of the doctor. Patients stable on methadone will be considered for participation.
* Have an active/acute CDC Category C event.
* Are unable to absorb or take medicines by mouth.
* Are pregnant or breast-feeding.
* Have a serious medical condition (such as diabetes, heart problem, hepatitis) that might affect the safety of the patient.
* Have had pancreatitis or hepatitis within the last 6 months.
* Have been treated with radiation or chemotherapy within 28 days before the study drug will be taken, or will have the need for these during the study.
* Have taken drugs that affect the immune system (such as corticosteroids, interleukins, interferons) or that have anti-HIV activity (such as hydroxyurea or foscarnet) within 28 days before the study drug will be taken.
* Have received HIV vaccine within 3 months before the study drug will be taken.
* Have received certain other drugs within 28 days before the study drug will be taken, or think that they will be needed during the study.
* Have received experimental treatments.
* Have allergies which might interfere with the study, in the opinion of the doctor.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 210
Dates: Start 2000-11

CONTACTS AND LOCATIONS:
Locations (23):
- United States (23):
  - East Bay Clinical Trial Ctr, Concord, California
  - Ocean View Internal Medicine, Long Beach, California
  - Florida ID Group, Orlando, Florida
  - Hillsborough County Health Dept, Tampa, Florida
  - Clinical Pharmacology Services, Tampa, Florida
  - Veterans Affairs Med Ctr of North Chicago, Chicago, Illinois
  - Univ of Kansas Med Ctr, Kansas City, Kansas
  - Saint Michael's Med Ctr, Newark, New Jersey
  - UMDNJ - New Jersey Med School, Newark, New Jersey
  - Addiction Research and Treatment Corp, Brooklyn, New York
  - Brookdale Univ Hosp and Med Ctr, Brooklyn, New York
  - Gervais Frechette, New York, New York
  - Howard Grossman, New York, New York
  - Mount Sinai School of Medicine, New York, New York
  - Univ of Rochester Med Ctr, Rochester, New York
  - Bronx Municipal Hosp Ctr/Jacobi Med Ctr, The Bronx, New York
  - SMO-USA Inc, Charlotte, North Carolina
  - Advanced Clinical Trials Inc, Eugene, Oregon
  - Thomas Jefferson Univ, Philadelphia, Pennsylvania
  - Univ of Texas Med Branch, Galveston, Texas
  - MacGregor Med Association, Houston, Texas
  - Walter Gaman, Irving, Texas
  - Southwest Texas Methodist Hosp, San Antonio, Texas